CLINICAL TRIAL: NCT06801548
Title: Fully Digital Guided Esthetic Crown Lengthening Surgery: Evaluation of Accuracy and Patient Satisfaction (A Randomized Controlled Clinical Study)
Brief Title: Fully Digital Guided Esthetic Crown Lengthening Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Abdallah Abdelnabi, Resident of Oral Medicine and Periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-ReclM122210
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-03

CONDITIONS: Gummy Smile
Keywords: Esthetic crown lengthening; Gingivectomy; Guided surgery; Wax-up; Digital

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional arm (Active Comparator): Esthetic crown lengthening surgery is done using mock-up based guide
  Interventions: Procedure: Esthetic crown lengthening surgery
- Digital arm (Active Comparator): Esthetic crown lengthening surgery is done using digital guide
  Interventions: Procedure: Esthetic crown lengthening surgery using Digital guide

INTERVENTIONS:
Procedure: Esthetic crown lengthening surgery — Esthetic crown lengthening surgery using mock-up based guide
  Arms: Conventional arm
Procedure: Esthetic crown lengthening surgery using Digital guide — Esthetic crown lengthening surgery using digital guide based on DSD and CBCT
  Arms: Digital arm

SUMMARY:
The goal of this randomized controlled clinical study is to compare Fully digital to wax-up/mock-up guided esthetic crown lengthening procedure in management of excessive gingival display caused by altered passive eruption type 1B

The main question it aims to answer is:

Does the fully digital guided gingivectomy approach able to introduce a more precise, accuracy and reliability technique with more patient satisfaction compared to the mock-up guided method?

DETAILED DESCRIPTION:
In today's world, the idea of smile and dental aesthetics extends beyond just the teeth. The fundamentals of a smile center on the interaction between the three key elements: the teeth, lips , and the gingiva.

Gummy smile (Excessive gingival display) is acknowledged by the American Academy of Periodontology (AAP) as a deformity and mucogingival problem that impacts the area surrounding the teeth

This condition may result from various etiological factors: short lip, hypermobile/hyperactive lip, short clinical crowns, dentoalveolar extrusion, altered passive eruption (APE), gingival hyperplasia, and vertical maxillary excess.

Altered passive eruption is described as "the gingival margin in adults is positioned incisal to the crown's cervical convexity and distanced from the tooth's cementoenamel junction."

Altered passive eruption defined as "the gingival margin in the adult is located incisal to the cervical convexity of the crown and removed from the cementoenamel junction of the tooth".

Altered passive eruption classified into two main classes according to the relationship of the gingiva to the anatomic crown and furthermore subdivided those classes according to the position of the osseous crest. The two types are subdivided into four categories: 1A, 1B and 2A, 2B.

The diagnosis of APE is made on a collective clinical and radiographic examination, it begins with analyzing the repose during a natural smile followed by analyzing the gingival display, the alveolar crest level, as well as the lip line of the patient.

Determination can be made whether a gingivectomy alone will suffice or a gingival flap will be needed with or without ostectomy will depend of the diagnosis of APE and classification of each case.

The selection of one technique over another depends on several patient related factors such as esthetics, clinical crown to root ratio, root proximity, root morphology, furcation location, individual tooth position, collective tooth position and ability to restore the teeth.

Esthetic crown lengthening (ECL) approach (both gingivectomy and bone removal) is used when less than 2 mm exists between the crest of the bone and the new gingival margin, and an adequate attached gingiva will remain after surgery (APE type IB).

Diagnostic mock-up fabricated using a temporary bis-acrylic resin with a putty guide directly from the wax-up can be used to provide the patient and clinician with an evaluation of the future outcome and can be used as a surgical guide for crown lengthening procedures.

The major limitations with wax-up/ mock-up guided esthetic crown lengthening procedure would be the time consumed during making and modifying conventional wax-ups as well as the unpredictable estimate of where the gingival margin should be.

Utilization of digital workflows allowed the enhancement of communication and might improve the predictability of contemporary ECL approach.

The introduction of computer-aided design and computer-aided manufacturing (CAD-CAM) techniques has helped surgeons perform more precise and predictable surgery and contributed to improved esthetics.

By combining the use of Digital Smile Design and CAD/CAM technology with (3D) printing, a surgical guide for ECL procedure could be produced.

The aim of the present study will be to evaluate accuracy and reliability of digital guided method of ECL procedure using CAD CAM technology versus conventional method using resin Mock-up as ECL surgical guide.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have Altered passive eruption (APE) type 1 B, according to classification of APE by Coslet et al.

Both genders aged from 20-50 years. Patients have thick gingival phenotype (thickness of gingiva is ≥ 1 mm) Patients should be systematically free from any disease.

Exclusion Criteria:

* Pregnant and lactating females.
* Heavy smoker ≥ 10 cigarettes/day.
* Poor oral hygiene.
* Patients with occlusal or malalignment problems.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Accuracy of both guides | Immediately after the surgery
  The accuracy can be measured by comparing the planned surgery and the actual result of the surgery Linear measurement in millimeters

SECONDARY OUTCOMES:
Patient satisfaction | 3 months after the surgery
  This can be measured using a questionnaire includes questions about patient expectations about the surgery, pain during and after the surgery, and the overall results
Marginal stability | 4 weeks and 3 months
  Gingival margin is been evaluated after 4 weeks and 3 months of the surgery using subsequent intraoral scanning Linear measurement in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E Amr, Ass.Prof, Study Director — Faculty of Dentistry - Ain Shams University
Locations (1):
- Faculty of Dentistry - Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vercruyssen M, Cox C, Coucke W, Naert I, Jacobs R, Quirynen M. A randomized clinical trial comparing guided implant surgery (bone- or mucosa-supported) with mental navigation or the use of a pilot-drill template. J Clin Periodontol. 2014 Jul;41(7):717-23. doi: 10.1111/jcpe.12231. Epub 2014 Apr 10. PMID 24460748
- [Background] Lee EA. Aesthetic crown lengthening: classification, biologic rationale, and treatment planning considerations. Pract Proced Aesthet Dent. 2004 Nov-Dec;16(10):769-78; quiz 780. PMID 15739921
- [Background] Ganji KK, Patil VA, John J. A Comparative Evaluation for Biologic Width following Surgical Crown Lengthening Using Gingivectomy and Ostectomy Procedure. Int J Dent. 2012;2012:479241. doi: 10.1155/2012/479241. Epub 2012 Aug 26. PMID 22969804
- [Background] Jepsen S, Caton JG, Albandar JM, Bissada NF, Bouchard P, Cortellini P, Demirel K, de Sanctis M, Ercoli C, Fan J, Geurs NC, Hughes FJ, Jin L, Kantarci A, Lalla E, Madianos PN, Matthews D, McGuire MK, Mills MP, Preshaw PM, Reynolds MA, Sculean A, Susin C, West NX, Yamazaki K. Periodontal manifestations of systemic diseases and developmental and acquired conditions: Consensus report of workgroup 3 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S237-S248. doi: 10.1002/JPER.17-0733. PMID 29926943
- [Background] Shobha KS, Mahantesha, Seshan H, Mani R, Kranti K. Clinical evaluation of the biological width following surgical crown-lengthening procedure: A prospective study. J Indian Soc Periodontol. 2010 Jul;14(3):160-7. doi: 10.4103/0972-124X.75910. PMID 21760669
- [Background] Nugala B, Kumar BS, Sahitya S, Krishna PM. Biologic width and its importance in periodontal and restorative dentistry. J Conserv Dent. 2012 Jan;15(1):12-7. doi: 10.4103/0972-0707.92599. PMID 22368328
- [Background] Liu X, Yu J, Zhou J, Tan J. A digitally guided dual technique for both gingival and bone resection during crown lengthening surgery. J Prosthet Dent. 2018 Mar;119(3):345-349. doi: 10.1016/j.prosdent.2017.04.018. Epub 2017 Jul 8. PMID 28689907
- [Background] Garber DA, Salama MA. The aesthetic smile: diagnosis and treatment. Periodontol 2000. 1996 Jun;11:18-28. doi: 10.1111/j.1600-0757.1996.tb00179.x. No abstract available. PMID 9567953
- [Background] Coslet JG, Vanarsdall R, Weisgold A. Diagnosis and classification of delayed passive eruption of the dentogingival junction in the adult. Alpha Omegan. 1977 Dec;70(3):24-8. No abstract available. PMID 276255
- [Background] Bhola M, Fairbairn PJ, Kolhatkar S, Chu SJ, Morris T, de Campos M. LipStaT: The Lip Stabilization Technique- Indications and Guidelines for Case Selection and Classification of Excessive Gingival Display. Int J Periodontics Restorative Dent. 2015 Jul-Aug;35(4):549-59. doi: 10.11607/prd.2059. PMID 26133145